CLINICAL TRIAL: NCT05350943
Title: Phase II Study to Evaluate the Efficacy and Safety of HAIC Combined With Toripalimab and Donafenib in Patients With Advanced Biliary Tract Cancer
Brief Title: HAIC Combined With Toripalimab and Donafenib for Advanced BTC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Lu Wang, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Lu Wang, MD, PhD, professor, Fudan University
Organization: Fudan University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-GZWK-04
Record Dates: First submitted 2022-03-24; First posted 2022-04-28 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Biliary Tract Adenocarcinoma
MeSH Terms: interventions — Gemcitabine; Oxaliplatin; toripalimab; donafenib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HAIC+Toripalimab+Donafenib (Experimental): HAIC(GEMOX)+Toripalimab+Donafenib
  Interventions: Procedure: HAIC; Drug: Gemcitabine; Drug: Oxaliplatin; Drug: Toripalimab; Drug: Donafenib

INTERVENTIONS:
Procedure: HAIC — After successful percutaneous hepatic artery cannulation, superior mesenteric arteriogram and hepatic arteriogram were performed, and after confirming that the subjects were eligible for enrollment according to the results, the hepatic artery was cannulated to the predetermined position. The catheter was connected to a syringe pump in the ward for continuous pumping of drugs.
Drug: Gemcitabine — 1000 mg/m^2 in 100ml saline solution IV, d1, Q3W
Drug: Oxaliplatin — 85 mg/m^2 in 500ml 5% glucose solution over 2 hours IV, d1, Q3W
Drug: Toripalimab — 3mg/kg (body weight < 60kg) or 240 mg（body weight>= 60kg）in 250 saline soluation, IV, Q3W
Drug: Donafenib — 0.2mg. P.O, BID, continuously

SUMMARY:
This is a single center, single arm, phase II, prospective study to evaluate the efficacy and safety of Hepatic Arterial Infusion Chemotherapy (HAIC) combined with PD-1 inhibitor immunotherapy Toripalimab and Tyrosine Kinase Inhibitor Donafenib in patients with advanced biliary tract cancer.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 80 years of age, of any sex;
* Histologically/Cytologically confirmed diagnosis of unresectable advanced adenocarcinoma of the gallbladder, intrahepatic bile duct and extrahepatic bile duct.
* At least one measurable lesion umder CT/MRI as defined by RECIST1.1 criteria
* Patients must have adequate organ and marrow function as defined below:

Blood test:

Hemoglobin (HB) ≥90 g/L Absolute neutrophil count (ANC) ≥1.5×10^9/L； Platelet (PLT) ≥80×10^9/L；

Biochemical test:

total bilirubin≤2×ULN (institutional upper limit of norm) AST(SGOT)/ALT(SGPT)≤2.5 ×ULN creatinine clearance≥ 50 ml/min as calculated by the Cockroft-Gault formula

* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score of 0-1;
* Indocyanine Green Retention Rates at 15 min (ICGR15<22%;
* Life expectancy of > 3 months;

Exclusion Criteria

* Patients with other malignant tumors should be excluded
* Female patients who are pregnant or breast-feeding. Female patients who are pregnant during the study should also exit.
* Patient has enter any other clinical trails within 4 weeks prior to study entry.
* Patient known with a severe and/or uncontrolled medical disease.
* Chronic non-healing wound/bone fracture
* History of organ transplant
* Patients with abnormal coagulation function (PT>16s, APTT>43s, TT>21s, Fbg<2g/L), those have bleeding tendency (14 days prior to randomization must meet: INR is within the normal range without any use of anticoagulants); patients treated with anticoagulants or vitamin K antagonists such as warfarin, heparin or analogous therapy; use for preventive purposes is permitted provided that the international normalized ratio of prothrombin time (INR) ≤ 1.5, take low-dose warfarin (1 mg PO, QD) or low-dose aspirin (do not exceed 100 mg per day);
* Previous history of aterial/venous thrombosis such as cerebrovascular accidents, pulmonary embolism or deep venous thrombosis within one year prior to patients recruitment.
* Hitstory of psychiatric drug abuse and hasn't come clean, or with psychiatric illness/social situations that would limit compliance with study requirements
* History of immunodeficiency, or other acquired/congenital immunodeficiency diseases
* Concomitant diseases that severely endanger the safety of the subject or affect the study completion according to the judgment of the investigator
* Willingness to sign a written informed consent document, with good compliance.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | through study completion, an average of 2 year
  the sum of complete response rate and partial response rate

SECONDARY OUTCOMES:
Disease Control rate (DCR) | through study completion, an average of 2 year
  the sum of complete response rate, partial response rate and stable disease rate
Progression-free survival (PFS) | through study completion, an average of 2 year
  Time from randomization to disease progression
Overall survival (OS) | through study completion, an average of 2 year
  Time from randomization to death for any cause
Number of participants with treatment-related adverse events as assessed by NCI CTCAE v4.0. | through study completion, an average of 2 year
  Unforeseen medical events occurred when the subjects received drug treatment or research, but there is not necessarily a causal relationship with the drugs used.
  Severe adverse events
Quality of life questionnaire | through study completion, an average of 2 year
  The concept of comprehensively evaluating the quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China